CLINICAL TRIAL: NCT05393921
Title: The Clinical Efficacy of Intravesical Botox Injections When Combined With HoLEP Surgery in Patients With Benign Prostatic Hyperplasia and Overactive Bladder
Brief Title: The Combined Effect of Intravesical Botox Injections and HoLEP Surgery in Treating Benign Prostatic Hyperplasia and Overactive Bladder
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of interest
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY20220495
Record Dates: First submitted 2022-05-20; First posted 2022-05-26 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Benign Prostatic Hyperplasia; Overactive Bladder
MeSH Terms: conditions — Prostatic Hyperplasia; Urinary Bladder, Overactive

STUDY DESIGN:
Intervention Model Description: This study will be a randomized clinical trial. The study team is interested in approaching and recruiting patients who were referred for HoLEP surgery for their urinary symptoms and also eligible for intravesical Botox injections. This cohort of patients will be recruited and randomized into two groups: a control group that would undergo HoLEP procedure only, and an experimental group that will undergo HoLEP procedure combined with an intravesical Botox injection.
  This study will utilize a 1:1 randomization scheme to assign participants to either the control group or the experimental group. Participants will not be blinded to the procedure they are receiving. No one on the study team including those involved in data analysis will be blinded to the study arm assignment. The investigators plan to recruit a maximum of 50 participants in each arm.
  The study's intervention is whether Botox injections are added during the surgery or not.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Patients receiving HoLEP surgery only (No Intervention): 50 patients diagnosed with benign prostatic hyperplasia and overactive bladder and referred for HoLEP to treat their urinary symptoms. No Botox injections will be given.
- Patients receiving HoLEP surgery + Intravesical Botox Injections (Experimental): 50 patients diagnosed with benign prostatic hyperplasia and overactive bladder and referred for HoLEP to treat their urinary symptoms. Botox injections will be given during the surgery.
  Interventions: Drug: Intravesical Botox injection

INTERVENTIONS:
Drug: Intravesical Botox injection — Intravesical botox injection given only in experimental group.100 units of Botox will be used and diluted in 10 mL of normal saline. 0.5 cc injections will be administered in 20 injection sites (trigone sparing).
  Arms: Patients receiving HoLEP surgery + Intravesical Botox Injections

SUMMARY:
Benign prostatic hyperplasia (BPH) is the most common benign neoplasm in men. Almost 90% of men in their 70s report lower urinary tract symptoms related to BPH. These symptoms carry a significant negative impact on the patients' quality of life.

Despite the wide availability of surgical offerings to relieve bladder outlet obstruction such as transurethral resection of the prostate (TURP), Holmium Laser Enucleation of the Prostate (HoLEP), and prostatectomy, many patients still suffer from persistent LUTS after undergoing these. A study describing postoperative outcomes following HoLEP revealed that patients with severe lower urinary tract symptoms, storage-positive sub-score, and high maximum urinary flow rate before the surgery were affected by a rebound of mainly storage symptoms 6-8 weeks after HoLEP and prolonged recovery from LUTS with 7.4% of them presenting for persistent urge complaints.

Optimizing the management approach for these patients has been limited by lack of high level evidence-based recommendations and expert consensus. Intravesical botox injections are well-established therapeutic options for several urinary disorders. The current practice offers intravesical botox injections to patients who suffer from persistent urinary symptoms few months after their BPH procedure. This study aims to evaluate if giving botox injections at the time of the HoLEP surgery would yield a better outcome than performing the two procedures separately at different times (few months apart).

The concomitant use of botox injection during bladder de-obstructing procedures has been previously studied in TURP and have showed a significant reduction of incontinence episodes and OAB symptoms in the group that were treated with botox injections after 36 weeks post TURP. This data may suggest promising potential of this intervention in managing persistent OAB symptoms in patients with BOO. However, the efficacy of combining HoLEP and bladder Botox injections has not been systematically studied and evaluated.

The aim of this study is to evaluate the effect of intravesical Botox injections on lower urinary tract symptoms (LUTS) when administered during HoLEP surgery in patients with bladder outlet obstruction (BOO) and overactive bladder symptoms (OAB). The investigators are interested in comparing the postoperative outcome in terms of recovery and symptom relief in patients who performed HoLEP surgery with bladder Botox injections versus those who performed HoLEP surgery only at 2 weeks,1 month, 3 months, and 6 months postoperatively.

The investigators hypothesize that administering bladder botox injections during HoLEP surgery is a combination treatment that will result in faster and more potent symptom relief compared to patients who received only a HoLEP surgery for their obstructive and irritative symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Males age > 40
* Patients diagnosed with Benign Prostatic Hyperplasia (BPH) and referred for HoLEP surgery
* Lower urinary tract symptoms (LUTS) of Overactive Bladder Syndrome (OABS) frequency - urgency - urge incontinence episodes - dysuria - nocturia and eligible for bladder botox injections
* International Prostate Symptom Score (IPSS) ≥ 17
* Overactive Bladder Symptom Score (OABSS) ≥ 7
* Participants have failed, are intolerant, or bad candidates for anticholinergic medication treatment for OAB

Exclusion Criteria:

* History of bladder/prostate cancer
* History of pelvic radiotherapy
* History of neurological diseases
* Presence of active Urinary Tract Infection (UTI)
* Previous Bladder Outlet Procedure (Transurethral resection of prostate (TURP) Transurethral Incision of Prostate (TUIP) - UroLift, etc..)
* History of adverse reaction to Botox injections
* Post-void residual (PVR) greater than 300 ml
* History of clean intermittent catheterization
* Patients unable to stop anticoagulation of antiplatelet inhibitors 3 days prior to procedure

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Change in International Prostate Symptom Score (IPSS) | IPSS scores will be recorded before the surgery and at 4 checkpoints after the surgery during every clinical visit: 2 weeks -1 month - 3 months - 6 months postoperatively
  Comparing the change in IPSS score between the two arms across time
Change in Overactive Bladder Symptoms Score (OABSS) | OABSS scores will be recorded before the surgery and at 4 checkpoints after the surgery during every clinical visit: 2 weeks -1 month - 3 months - 6 months postoperatively
  Comparing the change in OABSS score between the two arms across time
Change in Maximum Urinary Flow rate | Uroflowmetry will be performed before the surgery and at 4 checkpoints after the surgery during every clinical visit: 2 weeks -1 month - 3 months - 6 months postoperatively
  Comparing the change in maximum urinary flow rate(mL/sec) between the two arms across time
Change in Post-Void Residual (PVR) Volume | Postvoid residual volume (mL) will be performed before the surgery and at 4 checkpoints after the surgery during every clinical visit: 2 weeks -1 month - 3 months - 6 months postoperatively
  Comparing the change in postvoid residual volume (mL) between the two arms across time

SECONDARY OUTCOMES:
Adverse events | Adverse events will be monitored throughout the entire study duration (6 months after the surgery)
  Any adverse events in the context of readmissions, emergency department visits, and clinical visits will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Michael Zell, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (3):
- United States (3):
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - UH Brainard Medical Bldg, Lyndhurst, Ohio
  - UH Regional Hospitals - Richmond Campus, Richmond Heights, Ohio

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available

REFERENCES:
- [Background] Antunes AA, Srougi M, Coelho RF, de Campos Freire G. Botulinum toxin for the treatment of lower urinary tract symptoms due to benign prostatic hyperplasia. Nat Clin Pract Urol. 2007 Mar;4(3):155-60. doi: 10.1038/ncpuro0735. PMID 17347660
- [Background] Ahyai SA, Marik I, Ludwig TA, Becker A, Asdjodi S, Kluth L, Chun F, Fisch M, Schmid M. Super early detailed assessment of lower urinary tract symptoms after holmium laser enucleation of the prostate (HoLEP): a prospective study. World J Urol. 2020 Dec;38(12):3207-3217. doi: 10.1007/s00345-020-03126-x. Epub 2020 Feb 21. PMID 32086571
- [Background] Rapp DE, Lucioni A, Bales GT. Botulinum toxin injection: a review of injection principles and protocols. Int Braz J Urol. 2007 Mar-Apr;33(2):132-41. doi: 10.1590/s1677-55382007000200002. PMID 17488531
- [Background] Allameh F, Basiri A, Razzaghi M, Abedi AR, Fallah-Karkan M, Ghiasy S, Hosseininia SM, Montazeri S. Clinical Efficacy of Transurethral Resection of the Prostate Combined with Oral Anticholinergics or Botulinum Toxin - A Injection to Treat Benign Prostatic Hyperplasia with Overactive Bladder: A Case-Control Study. Clin Pharmacol. 2020 Jun 26;12:75-81. doi: 10.2147/CPAA.S256051. eCollection 2020. PMID 32617023
- [Background] Fusco F, Creta M, De Nunzio C, Iacovelli V, Mangiapia F, Li Marzi V, Finazzi Agro E. Progressive bladder remodeling due to bladder outlet obstruction: a systematic review of morphological and molecular evidences in humans. BMC Urol. 2018 Mar 9;18(1):15. doi: 10.1186/s12894-018-0329-4. PMID 29519236